CLINICAL TRIAL: NCT00940225
Title: A Randomized Discontinuation Study of XL184 in Subjects With Advanced Solid Tumors
Brief Title: Study of Cabozantinib (XL184) in Adults With Advanced Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-203
Record Dates: First submitted 2009-07-12; First posted 2009-07-15 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumors; Cancer
Keywords: Metastatic Breast Cancer (MBC); Melanoma; Stomach or Gastroesophageal Junction Carcinoma (GEJ); Hepatocellular Carcinoma (HCC); Small Cell Lung Cancer (SCLC); Non-Small Cell Lung Cancer (NSCLC); Ovarian Cancer; Pancreatic Cancer; Prostate Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Melanoma; Carcinoma, Hepatocellular; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Lead-in Stage - cabozantinib (XL184) (Experimental): Open Label, cabozantinib, 100 mg, po QD for 12 weeks.
  Interventions: Drug: Cabozantinib
- Randomized Stage - cabozantinib (XL184) (Experimental): Blinded, cabozantinib, 100 mg, po QD until disease progression.
  Interventions: Drug: Cabozantinib
- Randomized Stage - placebo (Placebo Comparator): Blinded, placebo, 100 mg, po QD until disease progression.
  Interventions: Drug: Placebo
- Open-Label Extension - cabozantinib (XL184) (Experimental): Open Label, cabozantinib, for subjects that were on placebo during the randomized stage, 100 mg, po QD until disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib
- Non-Randomized Expansion (NRE) Cohort - Castrate Resistant Prostate Cancer (CRPC), 100mg (Experimental): Open Label, cabozantinib, 100 mg, po QD until disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib
- Non-Randomized Expansion (NRE) Cohort - Castrate Resistant Prostate Cancer (CRPC), 39.4mg (Experimental): Open Label, cabozantinib, 39.4, po QD until disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib
- A. Non-Randomized Expansion (NRE) Cohort - Ovarian (Experimental): Open Label, cabozantinib, 100 mg, po QD until disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib
  Other Names: XL184
  Arms: A. Non-Randomized Expansion (NRE) Cohort - Ovarian; Lead-in Stage - cabozantinib (XL184); Non-Randomized Expansion (NRE) Cohort - Castrate Resistant Prostate Cancer (CRPC), 100mg; Non-Randomized Expansion (NRE) Cohort - Castrate Resistant Prostate Cancer (CRPC), 39.4mg; Open-Label Extension - cabozantinib (XL184); Randomized Stage - cabozantinib (XL184)
Drug: Placebo
  Arms: Randomized Stage - placebo

SUMMARY:
This is a Phase 2 study to evaluate the efficacy and safety of cabozantinib (XL184) in subjects with selected advanced tumor types.

DETAILED DESCRIPTION:
The goal of this clinical trial was to learn about the efficacy, safety, and tolerability of cabozantinib against a placebo in subjects with Metastatic Breast Cancer (MBC), Gastric and Gastroesophageal Junction Cancer (GEJ), Hepatocellular Carcinoma (HCC), Melanoma, Non-small Cell Lung Cancer (NSCLC), Ovarian (primary peritoneal or fallopian tube carcinoma), Pancreatic Cancer, Castration-Resistant Prostate Cancer (CRPC), or Small cell Lung Cancer (SCLC) with advanced tumors.

The main questions this study aimed to answer were:

* What is the efficacy of cabozantinib in subjects with advanced solid tumors?
* What is the safety and efficacy of cabozantinib at two starting dose levels 100 milligrams (mg) once daily (po QD) and 39.4 mg po QD? Please note: that the 39.4 mg, po QD was only used in the Non-Randomized Expansion (NRE) part of the study

There were three stages to the Randomized Discontinuation Trial (RDT):

1. The Lead in Stage: This stage enrolled eligible patients with advanced solid tumors who received open-label cabozantinib at 100 mg once daily for 12 weeks.
2. The Randomized Stage: Subjects who demonstrated stable disease (SD) at the end of 12 weeks of the Lead-in Stage were randomized to receive cabozantinib or placebo (a look-alike substance that contains no active drug) in a blinded manner.

   After randomization, when a patient developed progressive disease (PD), study treatments were discontinued and the treatment blind was broken. If the subject was on a placebo, the subject was offered the opportunity to receive cabozantinib. If the subject was already on cabozantinib, the subject entered the Post-Treatment Period where they were followed until death.
3. Open-Label Extension: Subjects who were deemed with partial response (PR) or complete response (CR) at Week 12 of the Lead-In Stage were not randomized but allowed to participate in the "Open Label Extension". Patients were given the cabozantinib treatment of 100 mg, po QD.

The emerging data supported enrollment in an open-label, Non-Randomized Expansion cohort (NRE). These cohorts targeted patients with prostate and ovarian cancers. For the patients with prostate, they were assigned to either 100 mg, po QD or 39.4 mg, po QD.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a cytologically or histologically and radiologically confirmed, advanced, recurrent, or metastatic solid tumor of the nine types listed below:

  * Pancreatic Cancer
  * Castration-Resistant Prostate Cancer (CRPC)
  * Hepatocellular Carcinoma (HCC)
  * Gastric or Gastroesophageal Junction Cancer
  * Melanoma
  * Small Cell Lung Cancer (SCLC)
  * Ovarian cancer, primary peritoneal or fallopian tube carcinoma
  * Breast cancer that is one of the following subtypes: estrogen receptor positive breast cancer, estrogen receptor/progesterone receptor/HER2-negative (triple-negative), or inflammatory (regardless of receptor status) disease histology
  * Non-Small Cell Lung Cancer (NSCLC)
* Certain requirements for prior therapies may apply
* The subject has documented progressive disease at screening
* Subjects having any tumor type of other than CRPC must have at least one lesion that is not within a previously irradiated field and is measurable on CT or MRI scan
* The subject has recovered to baseline or CTCAE ≤ Grade 1 from toxicities related to prior treatment (some exceptions apply)
* The subject is ≥ 18 years old on the day of consent
* Tissue samples from archival or fresh tissue, or a tissue block of the subject's tumor
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* The subject has adequate organ function
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Sexually active fertile subjects (male and female), and their partners, must agree to use medically accepted methods of contraception during the course of the study and for 3 months after the last dose of the study drug(s)
* Female subjects of childbearing potential must have a negative pregnancy test at screening

Exclusion Criteria:

* The subject has experienced clinically-significant hematemesis or hemoptysis of >0.5 teaspoon of red blood, or other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has a cavitating pulmonary lesion(s) or a pulmonary lesion abutting or encasing a major blood vessel
* Certain restrictions on prior treatments apply
* The subject has known symptomatic or uncontrolled brain metastases or epidural disease
* The subject has prothrombin time/International Normalized Ratio (PT/INR) or partial thromboplastin time (PTT) test results that are above (1.3x)the laboratory upper limit of normal
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or Coumadin-related agents, heparin, thrombin or FXa inhibitors, and antiplatelet agents (low-dose aspirin (≤81 mg/day), low-dose warfarin (≤1mg/day, and prophylactic low molecular weight heparin (LMWH) are permitted)
* The subject has a corrected QT interval(QTcF)>500 ms at screening
* The subject has uncontrolled, significant intercurrent illness
* The subject is unable to swallow capsules
* The subject is pregnant or breastfeeding
* The subject has a previously-identified allergy or hypersensitivity to components of the study treatment formulation
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had another diagnosis of malignancy requiring systemic treatment within the last two years, unless non-melanoma skin cancer, in-situ carcinoma of the cervix, or superficial bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (34):
  - Pinnacle Oncology of Arizona, Scottsdale, Arizona
  - University of California Davis Cancer Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Dana Farber Cancer Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - Kansas City Cancer Center, Lee's Summit, Missouri
  - Midwest Hematology Oncology Consultants, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University GYN Oncology, Hilliard, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Northwest Cancer Specialists, Tualatin, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, ITOR, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Texas, M. D., Anderson Cancer Center, Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Fairfax Northern Virginia Hematology Oncology, Fairfax, Virginia
  - University of Washington, Seattle, Washington
- Belgium (5):
  - One Study Location, Brussels
  - One Study Location, Jette
  - Multiple Study Locations, Leuven
  - Liège
  - One Study Location, Mons
- Israel (4):
  - One Study Location, Jerusalem
  - One Study Location, Tel Aviv
  - One Study Location, Tel Litwinsky
  - One Study Location, Ẕerifin
- Taiwan (3):
  - Multiple Study Locations, Tainan
  - Chang Gung Medical Foundation, Taoyuan County, Taipei
  - Taipei
- One Study Location, London, United Kingdom

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Schoffski P, Gordon M, Smith DC, Kurzrock R, Daud A, Vogelzang NJ, Lee Y, Scheffold C, Shapiro GI. Phase II randomised discontinuation trial of cabozantinib in patients with advanced solid tumours. Eur J Cancer. 2017 Nov;86:296-304. doi: 10.1016/j.ejca.2017.09.011. Epub 2017 Oct 20. PMID 29059635
- [Derived] Vergote IB, Smith DC, Berger R, Kurzrock R, Vogelzang NJ, Sella A, Wheler J, Lee Y, Foster PG, Weitzman R, Buckanovich RJ. A phase 2 randomised discontinuation trial of cabozantinib in patients with ovarian carcinoma. Eur J Cancer. 2017 Sep;83:229-236. doi: 10.1016/j.ejca.2017.06.018. Epub 2017 Jul 26. PMID 28755607
- [Derived] Kelley RK, Verslype C, Cohn AL, Yang TS, Su WC, Burris H, Braiteh F, Vogelzang N, Spira A, Foster P, Lee Y, Van Cutsem E. Cabozantinib in hepatocellular carcinoma: results of a phase 2 placebo-controlled randomized discontinuation study. Ann Oncol. 2017 Mar 1;28(3):528-534. doi: 10.1093/annonc/mdw651. PMID 28426123
- [Derived] Tolaney SM, Nechushtan H, Ron IG, Schoffski P, Awada A, Yasenchak CA, Laird AD, O'Keeffe B, Shapiro GI, Winer EP. Cabozantinib for metastatic breast carcinoma: results of a phase II placebo-controlled randomized discontinuation study. Breast Cancer Res Treat. 2016 Nov;160(2):305-312. doi: 10.1007/s10549-016-4001-y. Epub 2016 Oct 6. PMID 27714541
- [Derived] Leibowitz-Amit R, Pintilie M, Khoja L, Azad AA, Berger R, Laird AD, Aftab DT, Chi KN, Joshua AM. Changes in plasma biomarkers following treatment with cabozantinib in metastatic castration-resistant prostate cancer: a post hoc analysis of an extension cohort of a phase II trial. J Transl Med. 2016 Jan 13;14:12. doi: 10.1186/s12967-015-0747-y. PMID 26762579
- [Derived] Smith MR, Sweeney CJ, Corn PG, Rathkopf DE, Smith DC, Hussain M, George DJ, Higano CS, Harzstark AL, Sartor AO, Vogelzang NJ, Gordon MS, de Bono JS, Haas NB, Logothetis CJ, Elfiky A, Scheffold C, Laird AD, Schimmoller F, Basch EM, Scher HI. Cabozantinib in chemotherapy-pretreated metastatic castration-resistant prostate cancer: results of a phase II nonrandomized expansion study. J Clin Oncol. 2014 Oct 20;32(30):3391-9. doi: 10.1200/JCO.2013.54.5954. Epub 2014 Sep 15. PMID 25225437
- [Derived] Basch E, Autio KA, Smith MR, Bennett AV, Weitzman AL, Scheffold C, Sweeney C, Rathkopf DE, Smith DC, George DJ, Higano CS, Harzstark AL, Sartor AO, Gordon MS, Vogelzang NJ, de Bono JS, Haas NB, Corn PG, Schimmoller F, Scher HI. Effects of cabozantinib on pain and narcotic use in patients with castration-resistant prostate cancer: results from a phase 2 nonrandomized expansion cohort. Eur Urol. 2015 Feb;67(2):310-8. doi: 10.1016/j.eururo.2014.02.013. Epub 2014 Feb 20. PMID 24631409
- [Derived] Smith DC, Smith MR, Sweeney C, Elfiky AA, Logothetis C, Corn PG, Vogelzang NJ, Small EJ, Harzstark AL, Gordon MS, Vaishampayan UN, Haas NB, Spira AI, Lara PN Jr, Lin CC, Srinivas S, Sella A, Schoffski P, Scheffold C, Weitzman AL, Hussain M. Cabozantinib in patients with advanced prostate cancer: results of a phase II randomized discontinuation trial. J Clin Oncol. 2013 Feb 1;31(4):412-9. doi: 10.1200/JCO.2012.45.0494. Epub 2012 Nov 19. PMID 23169517

RESULTS

PARTICIPANT FLOW:
Groups:
- RDT Cohort - Castration-Resistant Prostate Cancer (CRPC); RDT Cohort - Melanoma; RDT Cohort - Non-Small Cell Lung Cancer (NSCLC); RDT Cohort - Pancreatic Cancer; RDT Cohort - Gastric/Gastroesophageal Junction Cancer (GEJ); RDT Cohort - Hepatocellular Carcinoma (HCC); RDT Cohort - Small Cell Lung Cancer (SCLC); RDT Cohort - Ovarian Cancer; RDT Cohort - Metastatic Breast Cancer (MBC): Eligible subjects with advanced solid tumors received open-label cabozantinib at a starting daily dose of 100 mg (freebase weight).
- NRE Cohort - CRPC 100 mg; NRE Cohort - Ovarian Cancer 100mg: Subjects received a single oral daily dose of cabozantinib at 100 mg.
- NRE Cohort - CRPC 39.4 mg: Subjects received a single oral daily dose of cabozantinib at 39.4 mg.
Period: Overall Study
Arm/Group | RDT Cohort - Castration-Resistant Prostate Cancer (CRPC) | RDT Cohort - Melanoma | RDT Cohort - Non-Small Cell Lung Cancer (NSCLC) | RDT Cohort - Pancreatic Cancer | RDT Cohort - Gastric/Gastroesophageal Junction Cancer (GEJ) | RDT Cohort - Hepatocellular Carcinoma (HCC) | RDT Cohort - Small Cell Lung Cancer (SCLC) | RDT Cohort - Ovarian Cancer | RDT Cohort - Metastatic Breast Cancer (MBC) | NRE Cohort - CRPC 100 mg | NRE Cohort - CRPC 39.4 mg | NRE Cohort - Ovarian Cancer 100mg
Started | 171 | 77 | 60 | 20 | 21 | 41 | 21 | 70 | 45 | 93 | 51 | 60
Completed | 156 | 66 | 47 | 16 | 19 | 36 | 20 | 60 | 41 | 87 | 48 | 54
Not Completed | 15 | 11 | 13 | 4 | 2 | 5 | 1 | 10 | 4 | 6 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- RDT Cohort - CRPC; RDT Cohort - Melanoma; RDT Cohort - NSCLC; RDT Cohort - Pancreatic Cancer; RDT Cohort - GEJ; RDT Cohort - HCC; RDT Cohort - SCLC; RDT Cohort - Ovarian Cancer; RDT Cohort - MBC: Eligible subjects with advanced solid tumors received open-label cabozantinib at a starting daily dose of 100 mg (freebase weight).
- Total: Total of all reporting groups
Arm/Group | RDT Cohort - CRPC | RDT Cohort - Melanoma | RDT Cohort - NSCLC | RDT Cohort - Pancreatic Cancer | RDT Cohort - GEJ | RDT Cohort - HCC | RDT Cohort - SCLC | RDT Cohort - Ovarian Cancer | RDT Cohort - MBC | NRE Cohort - CRPC 100 mg | NRE Cohort - CRPC 39.4 mg | NRE Cohort - Ovarian Cancer 100mg | Total
Number analyzed (Participants) | 171 | 77 | 60 | 20 | 21 | 41 | 21 | 70 | 45 | 93 | 51 | 60 | 730
Age, Customized [Count of Participants; unit: Participants]
  <= 40 years | 0 | 5 | 1 | 1 | 1 | 4 | 0 | 4 | 6 | 0 | 0 | 1 | 23
  > 40 - <= 50 years | 4 | 6 | 3 | 1 | 3 | 3 | 2 | 12 | 7 | 3 | 5 | 10 | 59
  > 50 - <= 65 years | 60 | 28 | 23 | 11 | 9 | 22 | 12 | 32 | 26 | 41 | 24 | 33 | 321
  > 65 years | 107 | 38 | 33 | 7 | 8 | 12 | 7 | 22 | 6 | 49 | 22 | 16 | 327
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 35 | 27 | 7 | 5 | 10 | 12 | 70 | 44 | 0 | 0 | 60 | 270
  Male | 171 | 42 | 33 | 13 | 16 | 31 | 9 | 0 | 1 | 93 | 51 | 0 | 460
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 2 | 2 | 0 | 1 | 15 | 1 | 0 | 1 | 1 | 1 | 4 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 11 | 2 | 6 | 2 | 1 | 3 | 1 | 0 | 1 | 4 | 2 | 2 | 35
  White | 145 | 72 | 51 | 18 | 19 | 22 | 18 | 66 | 41 | 85 | 45 | 51 | 633
  More than one race | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 9
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) - LEAD IN STAGE, RDT Cohorts and NRE Ovarian Cohort Only
Description: Objective response rate (ORR) per modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.0 per investigator
  The analysis of ORR in the RDT Cohorts were defined as the proportion of subjects with a best overall response of confirmed complete response (CR) or partial response (PR) per mRECIST 1.0 during the 12-week Lead-In Stage.
  In the NRE Ovarian Cohort, mRECIST 1.1 was used. ORR for the NRE CRPC Cohorts was not a primary objective and is therefore not captured in the table below.
Time Frame: From initial dose through final study visit up to 44 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Lead-in Stage - CRPC; Lead-in Stage - Melanoma; Lead-in Stage - NSCLC; Lead-in Stage - Pancreatic Cancer; Lead-in Stage - Gastric/GEJ; Lead-in Stage - Hepatocellular Carcinoma; Lead-in Stage - SCLC; Lead-in Stage - Ovarian Cancer; Lead-in Stage - Metastatic Breast Cancer; Lead-in Stage - NRE Ovarian Cancer: cabozantinib, 100 mg, po QD for 12 weeks
Arm/Group | Lead-in Stage - CRPC | Lead-in Stage - Melanoma | Lead-in Stage - NSCLC | Lead-in Stage - Pancreatic Cancer | Lead-in Stage - Gastric/GEJ | Lead-in Stage - Hepatocellular Carcinoma | Lead-in Stage - SCLC | Lead-in Stage - Ovarian Cancer | Lead-in Stage - Metastatic Breast Cancer | Lead-in Stage - NRE Ovarian Cancer
Number analyzed (Participants) | 171 | 77 | 60 | 20 | 21 | 41 | 21 | 70 | 45 | 60
percentage of participants | 4.7 [2.0 to 8.7] | 5.2 [1.8 to 12.4] | 10 [4.4 to 20.3] | 0 [0 to 15.4] | 4.8 [0.2 to 21.8] | 4.9 [0.9 to 16.1] | 4.8 [0.2 to 21.8] | 21.7 [13.1 to 32.4] | 13.6 [6.0 to 25.7] | 10.0 [3.3 to 21.8]

2. Primary Outcome: Bone Scan Response (BSR) - NRE, CRPC
Description: The reduction of bone scan lesion area (BSLA) by > 30% was used as the quantitative measure of BSR. BSR was a primary outcome measure for only the NRE CRPC Cohorts.
Time Frame: From initial dose through final study visit up to 15 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- NRE Cohort - CRPC 100 mg: cabozantinib, 100 milligrams orally, daily for 12 weeks until progression or unacceptable toxicity.
- NRE Cohort - CRPC 39.4 mg: cabozantinib, 39.4 milligrams orally, daily for 12 weeks until progression or unacceptable toxicity.
Arm/Group | NRE Cohort - CRPC 100 mg | NRE Cohort - CRPC 39.4 mg
Number analyzed (Participants) | 93 | 51
percentage of participants | 74.2 [64.1 to 82.7] | 47.1 [32.9 to 61.5]

3. Primary Outcome: Progression-Free Survival (PFS) - Randomized Stage, RDT Cohorts Only
Description: Progression Free Survival during the Randomized Stage (Randomized Population)
Time Frame: From initial dose through final study visit up to 44 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Randomized Phase - CRPC, Cabozantinib Arm; Randomized Phase - Melanoma, Cabozantinib Arm; Randomized Phase - NSCLC, Cabozantinib Arm; Randomized Phase - Pancreatic Cancer, Cabozantinib Arm; Randomized Phase - Gastric/GEJ, Cabozantinib Arm; Randomized Phase - HCC, Cabozantinib Arm; Randomized Phase - SCLC, Cabozantinib Arm; Randomized Phase - Ovarian Cancer, Cabozantinib Arm; Randomized Phase - MBC, Cabozantinib Arm: cabozantinib, 100 mg, po QD, ongoing until progression
- Randomized Phase - CRPC, Placebo Arm: placebo 100mg, po QD, ongoing until progression
- Randomized Phase - Melanoma, Placebo Arm; Randomized Phase - NSCLC, Placebo Arm; Randomized Phase - Pancreatic Cancer, Placebo Arm; Randomized Phase - Gastric/GEJ , Placebo Arm: Placebo, 100mg, po QD, ongoing until progression
- Randomized Phase - HCC, Placebo Arm; Randomized Phase - SCLC, Placebo Arm; Randomized Phase - Ovarian Cancer, Placebo Arm; Randomized Phase - MBC, Placebo Arm: placebo, 100 mg, po QD, ongoing until progression
Arm/Group | Randomized Phase - CRPC, Cabozantinib Arm | Randomized Phase - CRPC, Placebo Arm | Randomized Phase - Melanoma, Cabozantinib Arm | Randomized Phase - Melanoma, Placebo Arm | Randomized Phase - NSCLC, Cabozantinib Arm | Randomized Phase - NSCLC, Placebo Arm | Randomized Phase - Pancreatic Cancer, Cabozantinib Arm | Randomized Phase - Pancreatic Cancer, Placebo Arm | Randomized Phase - Gastric/GEJ, Cabozantinib Arm | Randomized Phase - Gastric/GEJ , Placebo Arm | Randomized Phase - HCC, Cabozantinib Arm | Randomized Phase - HCC, Placebo Arm | Randomized Phase - SCLC, Cabozantinib Arm | Randomized Phase - SCLC, Placebo Arm | Randomized Phase - Ovarian Cancer, Cabozantinib Arm | Randomized Phase - Ovarian Cancer, Placebo Arm | Randomized Phase - MBC, Cabozantinib Arm | Randomized Phase - MBC, Placebo Arm
Number analyzed (Participants) | 14 | 17 | 13 | 13 | 8 | 8 | 3 | 3 | 3 | 2 | 10 | 12 | 8 | 2 | 7 | 6 | 5 | 5
months | 5.5 [4.0 to 8.5] | 1.4 [1.25 to 2.73] | 4.5 [1.8 to 15.4] | 2.8 [1.45 to 5.45] | 2.4 [1.3 to 2.9] | 2.4 [1.4 to 2.7] | 2.8 [1.5 to 2.8] | .07 [.07 to .07] | NA [2.3 to NA] — There was only one out of three subjects evaluated; unable to estimate due to insufficient number of patients within cohort. | 1.0 [.72 to 1.38] | 2.5 [1.3 to 6.8] | 1.4 [1.3 to 4.2] | 5.5 [1.9 to 6.9] | 1.5 [.85 to 2.23] | 4.9 [3.9 to 13.6] | 1.4 [1.3 to 1.6] | 6.9 [5.1 to 13.5] | 1.1 [.7 to 1.3]

4. Secondary Outcome: Duration of Objective Response (OR) - Responders From Lead-in Stage
Description: Duration of objective response was defined as the time from the tumor assessment that first documented PR or CR that was subsequently confirmed at least 28 days later until the date of documented progression. There were either few or no responders in the Gastric/GEJ, SCLC, and pancreatic cohorts so these cohorts are excluded.
Time Frame: From initial dose through final study visit up to 44 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- CRPC; Melanoma; NSCLC; Hepatocellular Carcinoma; Ovarian Cancer; Metastatic Breast Cancer: cabozantinib, 100 mg, po QD ongoing until progression
Arm/Group | CRPC | Melanoma | NSCLC | Hepatocellular Carcinoma | Ovarian Cancer | Metastatic Breast Cancer
Number analyzed (Participants) | 15 | 6 | 6 | 3 | 15 | 6
Months | 5.59 [4.27 to 8.34] | 5.55 [2.99 to 13.86] | 6.90 [5.29 to 10.74] | 4.21 [2.99 to NA] — Unable to estimate due to low numbers. | 11.24 [7.20 to NA] — Unable to estimate due to low numbers. | 3.29 [2.79 to 4.21]

5. Secondary Outcome: Progression Free Survival (PFS) - Throughout the Study
Description: Progression-free survival (PFS) from first dose throughout the study was estimated for all subjects (safety population) using a piecewise method.
Time Frame: From initial dose through final study visit up to 44 months
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- CRPC; Melanoma; NSCL; Pancreatic Cancer; Gastric/GEJ; Hepatocellular Carcinoma; SCLC; Ovarian Cancer; Metastatic Breast Cancer: cabozantinib, 100 mg, po QD
Arm/Group | CRPC | Melanoma | NSCL | Pancreatic Cancer | Gastric/GEJ | Hepatocellular Carcinoma | SCLC | Ovarian Cancer | Metastatic Breast Cancer
Number analyzed (Participants) | 171 | 77 | 60 | 20 | 21 | 41 | 21 | 70 | 45
months | 6.8 [3.9 to 9.7] | 2.8 [1.4 to 6.9] | 4.0 [1.4 to 5.7] | 2.7 [1.3 to 5.5] | 1.4 [1.3 to NA] — Unable to estimate as number of events is too low. | 5.2 [3.6 to 9.3] | 3.4 [1.4 to 8.2] | 5.5 [2.7 to 11.0] | 4.3 [1.4 to 8.1]

6. Secondary Outcome: Duration of Bone Scan Response - NRE Cohorts, CRPC Only
Description: The duration of BSR per IRF was calculated for CRPC subjects with an objective response (CR or PR) during the study.
Time Frame: From initial dose through final study visit up to 15 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- NRE Cohort - CRPC 100 mg: cabozantinib, 100 milligrams po QD for 12 weeks until progression or unacceptable toxicity.
- NRE Cohort - CRPC 39.4 mg: cabozantinib, 39.4 milligrams po QD for 12 weeks until progression or unacceptable toxicity.
Arm/Group | NRE Cohort - CRPC 100 mg | NRE Cohort - CRPC 39.4 mg
Number analyzed (Participants) | 69 | 24
months | 5.2 [4.07 to 6.67] | NA [NA to NA] — Unable to Estimate due to low numbers.

7. Secondary Outcome: Overall Survival (OS) - NRE Cohorts, CRPC and Ovarian Only
Time Frame: From initial dose through final study visit up to 15 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- NRE Cohort - Ovarian 100 mg: cabozantinib, 100 milligrams orally, daily for 12 weeks until progression or unacceptable toxicity.
Arm/Group | NRE Cohort - CRPC 100 mg | NRE Cohort - CRPC 39.4 mg | NRE Cohort - Ovarian 100 mg
Number analyzed (Participants) | 93 | 51 | 60
months | 11.1 [9.17 to 13.34] | 8.0 [7.92 to NA] — Unable to Estimate due to low numbers. | 8.5 [5.88 to 11.73]

ADVERSE EVENTS:
Groups:
- RDT All Cohorts: Includes all tumor types from the 203 RDT cohort: castration-resistant prostate cancer (CRPC), melanoma, non-small cell lung cancer (NSCLC), pancreatic cancer, gastric/gastroesophageal junction (GEJ) cancer, hepatocellular carcinoma (HCC), small cell lung cancer (SCLC), ovarian cancer, and metastatic breast cancer
- NRE Cohort - CRPC 100mg (Castration-Resistant Prostate Cancer); NRE Cohort - Ovarian 100mg: Subjects received a single oral daily dose of cabozantinib at 100 mg.
- NRE Cohort - CRPC 39.4mg (Castration-Resistant Prostate Cancer): Subjects received a single oral daily dose of cabozantinib at 39.4 mg.
Arm/Group | RDT All Cohorts | NRE Cohort - CRPC 100mg (Castration-Resistant Prostate Cancer) | NRE Cohort - CRPC 39.4mg (Castration-Resistant Prostate Cancer) | NRE Cohort - Ovarian 100mg
All-Cause Mortality (participants affected / at risk) | 54/526 | 53/93 | 13/51 | 33/60
Serious Adverse Events (participants affected / at risk) | 223/526 | 53/93 | 30/51 | 34/60
Other Adverse Events (participants affected / at risk) | 524/526 | 93/93 | 50/51 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RDT All Cohorts (N=526) | NRE Cohort - CRPC 100mg (Castration-Resistant Prostate Cancer) (N=93) | NRE Cohort - CRPC 39.4mg (Castration-Resistant Prostate Cancer) (N=51) | NRE Cohort - Ovarian 100mg (N=60)
Anaemia (Blood and lymphatic system disorders) | 8 | 4 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 4 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 2 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 1 | 0
Atrioventricular Block (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 9 | 2 | 2 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 15 | 2 | 0 | 3
Diverticular Perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0 | 0 | 4
Intestinal Perforation (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 12 | 9 | 0 | 8
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritoneal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal Stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 5 | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 15 | 7 | 0 | 11
Asthenia (General disorders) | 9 | 1 | 1 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Drug Withdrawal Syndrome (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 1 | 1
General Physical Health Deterioration (General disorders) | 5 | 0 | 0 | 3
Malaise (General disorders) | 1 | 0 | 0 | 0
Multi-Organ Failure (General disorders) | 4 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 3 | 0 | 0 | 0
Pain (General disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 2 | 0 | 4
Acute Hepatic Failure (General disorders) | 1 | 0 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 5 | 1 | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Douglas' Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia Bacteremia (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0
Herpes Oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 1 | 0 | 0
Pelvic Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 16 | 3 | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 5 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 2 | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 5 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0
Wound Infection (Infections and infestations) | 2 | 0 | 0 | 0
Wound Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation Pneumonitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Amylase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 1
Blood Uric Acid Increased (Investigations) | 1 | 0 | 0 | 0
Lipase Increased (Investigations) | 1 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 17 | 6 | 2 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 2 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 4 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intracranial Tumor Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Squamous Cell Carcinoma of the Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 2 | 0 | 0 | 0
Occipital Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Speech Disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 1 | 1 | 0
Subdural Effusion (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 3 | 1 | 0 | 0
VIth Nerve Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 6 | 2 | 0 | 1
Mental Status Change (Psychiatric disorders) | 9 | 0 | 0 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 0
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 1 | 1 | 0
Renal Failure (Renal and urinary disorders) | 5 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 11 | 4 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urethral Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 23 | 7 | 8 | 1
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 12 | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 5 | 1 | 0 | 0
Hypovolaemic Shock (Vascular disorders) | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Pelvic Venous Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous Stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Corneal Epithelium Defect (Eye disorders) | 0 | 0 | 0 | 1
Macular Oedema (Eye disorders) | 0 | 1 | 0 | 0
Parophthalmia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal Hematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Performance Status Decreased (General disorders) | 0 | 0 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0
Diabetic Foot Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1
Blood Sodium Decreased (Investigations) | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bleeding Varicose Vein (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RDT All Cohorts (N=526) | NRE Cohort - CRPC 100mg (Castration-Resistant Prostate Cancer) (N=93) | NRE Cohort - CRPC 39.4mg (Castration-Resistant Prostate Cancer) (N=51) | NRE Cohort - Ovarian 100mg (N=60)
Anaemia (Blood and lymphatic system disorders) | 63 | 29 | 5 | 10
Leukopenia (Blood and lymphatic system disorders) | 27 | 7 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 35 | 8 | 3 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 58 | 10 | 3 | 9
Hypothyroidism (Endocrine disorders) | 66 | 30 | 4 | 15
Abdominal Distension (Gastrointestinal disorders) | 31 | 4 | 3 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 52 | 6 | 3 | 7
Constipation (Gastrointestinal disorders) | 168 | 32 | 16 | 21
Diarrhoea (Gastrointestinal disorders) | 314 | 66 | 23 | 46
Dry Mouth (Gastrointestinal disorders) | 87 | 9 | 4 | 12
Dyspepsia (Gastrointestinal disorders) | 63 | 12 | 7 | 15
Dysphagia (Gastrointestinal disorders) | 38 | 5 | 0 | 8
Flatulence (Gastrointestinal disorders) | 33 | 8 | 3 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 45 | 6 | 5 | 9
Glossodynia (Gastrointestinal disorders) | 42 | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 269 | 64 | 30 | 36
Oral Pain (Gastrointestinal disorders) | 68 | 11 | 2 | 4
Stomatitis (Gastrointestinal disorders) | 99 | 15 | 5 | 17
Vomiting (Gastrointestinal disorders) | 188 | 38 | 19 | 25
Asthenia (General disorders) | 115 | 18 | 7 | 10
Fatigue (General disorders) | 345 | 76 | 32 | 47
Mucosal Inflammation (General disorders) | 84 | 14 | 8 | 10
Oedema Peripheral (General disorders) | 76 | 13 | 11 | 7
Pain (General disorders) | 36 | 5 | 6 | 4
Pyrexia (General disorders) | 47 | 6 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 59 | 5 | 4 | 11
Alanine Aminotransferase Increased (Investigations) | 71 | 7 | 3 | 16
Aspartate Aminotransferase Increased (Investigations) | 94 | 10 | 5 | 21
Lipase Increased (Investigations) | 35 | 2 | 1 | 3
Weight Decreased (Investigations) | 165 | 42 | 19 | 18
Decreased Appetite (Metabolism and nutrition disorders) | 270 | 70 | 22 | 31
Dehydration (Metabolism and nutrition disorders) | 74 | 17 | 3 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 62 | 14 | 6 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 70 | 6 | 3 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 6 | 3 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 41 | 5 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 29 | 6 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 74 | 30 | 11 | 10
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 56 | 10 | 9 | 13
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 27 | 13 | 3 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 34 | 21 | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 36 | 9 | 1 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 90 | 29 | 11 | 9
Dizziness (Nervous system disorders) | 86 | 15 | 7 | 18
Dysgeusia (Nervous system disorders) | 156 | 35 | 14 | 21
Headache (Nervous system disorders) | 79 | 13 | 8 | 17
Neuropathy Peripheral (Nervous system disorders) | 38 | 7 | 0 | 6
Anxiety (Psychiatric disorders) | 34 | 2 | 1 | 8
Confusional State (Psychiatric disorders) | 35 | 7 | 0 | 2
Depression (Psychiatric disorders) | 38 | 4 | 2 | 4
Insomnia (Psychiatric disorders) | 44 | 7 | 2 | 4
Dysuria (Renal and urinary disorders) | 27 | 3 | 4 | 4
Proteinuria (Renal and urinary disorders) | 34 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 88 | 14 | 3 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 142 | 34 | 9 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 102 | 29 | 12 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 | 7 | 1 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 60 | 3 | 4 | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 23 | 7 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 1 | 0 | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 54 | 6 | 4 | 7
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 53 | 4 | 0 | 8
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 179 | 24 | 7 | 20
Rash (Skin and subcutaneous tissue disorders) | 102 | 19 | 6 | 12
Hypertension (Vascular disorders) | 126 | 25 | 10 | 19
Abdominal Pain (Gastrointestinal disorders) | 120 | 17 | 8 | 23
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 12 | 6 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 13 | 6 | 0
Hypotension (Vascular disorders) | 0 | 10 | 2 | 1
Chest Pain (Gastrointestinal disorders) | 0 | 8 | 3 | 2
Pallor (Vascular disorders) | 0 | 7 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 5 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 6 | 2 | 5
Platelet Count Decreased (Investigations) | 0 | 5 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 6 | 3 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 5 | 1 | 0
Chills (General disorders) | 0 | 5 | 0 | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 3 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 5 | 2 | 0
Hot Flush (Vascular disorders) | 0 | 5 | 0 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 5 | 2 | 2
Spinal Pain (General disorders) | 0 | 5 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 4 | 3 | 2
Haematuria (Renal and urinary disorders) | 0 | 3 | 6 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 10
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 5 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 4
Transaminases Increased (Investigations) | 0 | 3 | 0 | 3
Urinary Incontinence (Renal and urinary disorders) | 0 | 3 | 4 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 3 | 11
Blood Creatinine Increased (Investigations) | 0 | 2 | 3 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 1 | 7
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Syncope (Nervous system disorders) | 0 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 2 | 1 | 3
Vision Blurred (Eye disorders) | 0 | 2 | 4 | 2
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 1 | 0 | 4
Chest Discomfort (General disorders) | 0 | 1 | 3 | 3
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 2 | 3
Dry Eye (Eye disorders) | 0 | 1 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 7
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 4
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 3
Early Satiety (Gastrointestinal disorders) | 0 | 0 | 1 | 3
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 5
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 0 | 3
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 3
Memory Impairment (Nervous system disorders) | 0 | 2 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes